CLINICAL TRIAL: NCT06421311
Title: Ambispective Observational Study of Muscle Invasive Urothelial Carcinoma Patients Treated With Adjuvant Nivolumab in France
Brief Title: Observational Study of Muscle Invasive Urothelial Carcinoma Participants Treated With Adjuvant Nivolumab in France
Acronym: URADJ
Status: Terminated | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1416
Record Dates: First submitted 2024-05-02; First posted 2024-05-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants with muscle invasive urothelial carcinoma receiving nivolumab
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab — According to approved product label (France)

SUMMARY:
This study will estimate the real-world effectiveness of adjuvant nivolumab therapy in adult participants with muscle invasive urothelial carcinoma (MIUC) in France.

ELIGIBILITY:
Inclusion Criteria:

* Participants with pathological evidence of muscle invasive urothelial carcinoma (originating in bladder, ureter, or renal pelvis) at high risk of recurrence after radical resection with programmed death-ligand 1 (PD-L1) tumour cell expression ≥ 1%:

  * Who received neoadjuvant chemotherapy OR
  * Who did not receive neoadjuvant chemotherapy and who are not eligible or refusing adjuvant cisplatin chemotherapy
* At least 18 years of age at the time of treatment decision
* Decision to treat with adjuvant nivolumab therapy has already been taken
* Participants who provide oral informed consent to participate in the study (or who express non-opposition to data collection during their lifetime for deceased patients enrolled retrospectively)

Exclusion Criteria:

* Participants with a current primary diagnosis of a cancer other than muscle invasive urothelial carcinoma within the past 5 years, ie, a cancer other than urothelial carcinoma that requires systemic or other treatment or has not been treated curatively (as per discretion of the investigator)
* Participants currently enrolled in an interventional clinical trial for their urothelial carcinoma. Patients who have completed their participation in an interventional trial or who are not receiving study drug anymore and who are only followed-up for overall survival (OS) can be enrolled. Patients enrolled in a clinical trial not evaluating an investigational drug can be enrolled (e.g. trial investigating novel imaging modalities).
* Pregnant women
* Participants under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants in France with muscle invasive urothelial carcinoma (MIUC) that have been prescribed adjuvant nivolumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) of participants | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60

SECONDARY OUTCOMES:
Time to recurrence (TRR) | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Distance metastases-free survival (DMFS) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Non-urothelial tract recurrence free survival (NUTRFS) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Locoregional disease free survival (LRFDS) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Overall survival (OS) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Disease specific survival (DSS) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Second progression-free survival (PFS2) | At months 3, 6, 9, 12, 18, 24, 30, 26, 48 and 60
Participant demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant history of other cancer(s | Baseline
Participant comorbidities pre-existing at the time of adjuvant therapy initiation | Index date
Participant renal function at treatment initiation | Day 1
Participant concomitant systemic treatment(s) | Day 1 and at months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Diagnosis of muscle-invasive urothelial carcinoma diagnosis | Baseline
Systemic neoadjuvant treatment history | Baseline
Surgery for muscle-invasive urothelial carcinoma | Baseline
Participant history of previous urothelial carcinoma | Baseline
PD-L1 status testing results | Baseline
Participant muscle Invasive urothelial carcinoma disease characteristics | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Time from initial diagnosis of muscle invasive disease to adjuvant treatment initiation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Delay in adjuvant nivolumab treatment initiation related to post-operative complications | Baseline
Time from radical surgery to adjuvant nivolumab treatment initiation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Adjuvant nivolumab treatment duration | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Number of adjuvant nivolumab treatment cycles | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Dose adjuvant nivolumab per cycle | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Reason for adjuvant nivolumab treatment interruption | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Reason for adjuvant nivolumab treatment discontinuation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Non-systemic treatments prescribed post adjuvant nivolumab discontinuation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Systemic treatment prescribed post adjuvant nivolumab discontinuation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Participant response to prescribed systemic treatment post adjuvant nivolumab discontinuation | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Participant adverse events | At months 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60
Participant reported outcomes as assessed by European Quality of Life-5 Dimensions (EQ-5D) Questionnaire | Baseline, and at months 3, 6, 9, 12, 18, 24, 30, and 36
  Prospective participants only

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts